CLINICAL TRIAL: NCT02118194
Title: Assessment of Home/Work Simulation Tasks and Community Mobility Skills in the ReWalk Powered Exoskeleton in Persons With Spinal Cord Injury
Brief Title: Home/Work, Community Mobility Skills in the ReWalk Exoskeleton in Persons With SCI
Acronym: VA_ReWalk2
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann M. Spungen, EdD, Research Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: JJPVAMC ReWalk2
Record Dates: First submitted 2014-03-28; First posted 2014-04-21 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: paraplegia; paralysis; robotics; walking; immobilization
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paraplegia, spinal cord injury: An exoskeleton-assisted walking system for people with paralysis from spinal cord injury at thoracic level 1 and below (paraplegia) will be used.

SUMMARY:
The overall goal of this project is to determine if non-ambulatory persons with spinal cord injury (SCI) who have already participated in at least 20 sessions of ReWalk training can be further trained to achieve more advanced skills for use in the home or work place environments and outdoor community mobility skills in the ReWalk exoskeleton.

DETAILED DESCRIPTION:
Evaluation criteria will consist of the level of assistance, number of sessions and time to perform each of the tasks. Because some of these tasks have never been performed in an exoskeleton there is no standardized information to set a goal. As such, level of assistance and time to complete those tasks will be recorded in each participant for a descriptive analysis. Other tests, such as the six-minute walk test (6mWT), 10 meter walk test (10mWT) and timed up and go (TUG) have a range of specific timed values that have been measured in the exoskeleton by our investigators and others. These exoskeletal-assisted walking tests have standardized criteria on which the participants will be evaluated.

Participants will attend three to four, one to two-hour sessions per week for a total of 20 sessions in six weeks. Each session will consist of exoskeletal-assisted skill practice during standing and walking mobility training. In order to determine the number of session to learn the tasks, measurements will be performed one time weekly for the task-specific skills and walking tests and again at the end of 20 sessions.

Participants will tested in the exoskeleton for ability to perform certain task-specific indoor and outdoor mobility skills.

Advanced indoor skills include, but are not limited to:

1. Performance on a an indoor six-minute walk test (6minWT) and ten meter walk test (10mWT) on a smooth floor and on carpet;
2. Timed up and go test (TUG) performance indoors on a smooth floor and on carpet;
3. Home/work skills include: manipulating items on a counter top, retrieving an item from an overhead cabinet, and/or retrieving an object from a refrigerator;
4. Door navigation skills include: a push button door, revolving door and/or a non-powered door;
5. Elevator Skills include: pressing the call button outside an elevator, navigate the elevator doors, pressing the floor selection buttons in an elevator, and/or exiting the elevator doors; and
6. Exoskeletal-assisted stair ascent and descent.

Advanced outdoor skills include, but are not limited to:

1. 10 mWT and 6minWT performance outdoors on concrete, asphalt, uneven surfaces, and grass.
2. Exoskeletal-assisted walking on incline slopes (assessed as time to navigate a specified distance) for: up slight slope, down slight slope, navigate up curb cut-out, and/or navigate down curb cut-out.
3. Ability to navigate up and/or down a curb (assessed as level of assistance required).

Note: Additional skills may be tested and recorded as per each individual's ability and competency.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with spinal cord injury (SCI) who have already participated in at least 20 ReWalk training sessions.

Exclusion Criteria:

1. Diagnosis of neurological injury other than SCI including: Multiple sclerosis (MS), Stroke, Cerebral Palsy (CP), Amyotrophic lateral sclerosis (ALS), Traumatic Brain injury (TBI), Spina bifida, Parkinson's disease (PD), or other neurological condition that the study physician considers in his/her clinical judgment to be exclusionary;
2. Severe concurrent medical disease, illness or condition;
3. Unhealed fractures;
4. Systemic or peripheral infection;
5. Atherosclerosis, congestive heart failure, or history of myocardial infarction;
6. Trunk and/or lower extremity pressure ulcers;
7. Other illness, that the study physician considers in his/her clinical judgment to be exclusionary;
8. Severe spasticity (defined by an Ashworth score of >4.0 or clinical impression of the study physician or physical therapist);
9. Significant contractures or heterotropic ossification of the lower extremities that prevent flexion and extension of the joint;
10. Distal femur and/or proximal tibia bone mineral density less than 0.59 cm2.
11. Femoral neck or the total proximal femur bone mineral density T-scores < -3.5;
12. Psychopathology documentation in the medical record or history of that may conflict with study objectives;
13. Hypertension (Systolic Blood Pressure >140, Diastolic Blood Pressure >90); and/or
14. Pregnancy and/or lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females with paraplegia (T1 and below) who are unable to walk on their own will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2022-10-06 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Number of sessions and level of assistance to achieve the advanced indoor and outdoor exoskeletal-assisted walking skills | Assessments are weekly during the 20-session protocol and at the end over a 6 week period
  The walking tests (10mWT, 6-minWT, TUG) will be performed indoors on tile/linoleum and carpet and outdoors on concrete, asphalt, grass, dirt, uneven surfaces, curbs, curb cutouts, and ramps.

SECONDARY OUTCOMES:
Number of sessions and level of assistance to achieve specific advanced indoor standing and door navigation skills | Assessments are weekly during the 20-session protocol and at the end over a 6 week period
  The advanced indoor standing skills include counter top work, retrieving of items from an overhead cabinet and from a refrigerator. The door navigation skills include a push button door, elevator doors, revolving doors, and non-powered doors.

OTHER OUTCOMES:
Number of sessions and level of assistance to achieve exoskeletal-assisted stair ascent and descent | Assessments are weekly during the 20-session protocol an at the end over a 6 week period
  Participants will be timed to ascend and descend 13 steps in a stair well.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Spungen, EdD, Principal Investigator — James J Peters VA Medical Center
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Yang A, Asselin P, Knezevic S, Kornfeld S, Spungen AM. Assessment of In-Hospital Walking Velocity and Level of Assistance in a Powered Exoskeleton in Persons with Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):100-9. doi: 10.1310/sci2102-100. Epub 2015 Apr 12. PMID 26364279
- See also: Spinal Cord Damage Research Center website — http://www.scirc.org